CLINICAL TRIAL: NCT05317143
Title: Evaluation of Prostate Cancer Margins
Status: Completed | Type: Observational
Sponsor: Intuitive Surgical (Industry)
Responsible Party: Sponsor
Other Study IDs: 1091459C
Record Dates: First submitted 2022-02-02; First posted 2022-04-07 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: None Retained — Prostate
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Evaluation of prostate cancer margins — Evaluation of prostate cancer margins

SUMMARY:
Pathological assessment of prostate tissue

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with prostate cancer
* Subject must be scheduled for robotic-assisted radical prostatectomy at the clinical site.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with prostate cancer who undergo robotic-assisted prostatectomy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-02-22 (Actual); Primary Completion 2022-11-10 (Actual); Study Completion 2022-11-10 (Actual)

PRIMARY OUTCOMES:
Positive Margin | Immediately postoperatively, expected same day as surgery
  Detection of positive margin

CONTACTS AND LOCATIONS:
Overall Officials: Jörn Hinrich Witt, PD Dr. med, Principal Investigator — St. Antonius, Hospital, Prostatazentrum Nordwest, Möllenweg 22, 48599 Gronau, Germany; Sami-Ramzi Leyh-Bannurah, PD Dr. med, Principal Investigator — St. Antonius, Hospital, Prostatazentrum Nordwest, Möllenweg 22, 48599 Gronau, Germany
Locations (1):
- St. Antonius Hospital, Prostatazentrum Nordwest, Gronau, Germany

IPD SHARING:
Plan to Share IPD: No